CLINICAL TRIAL: NCT03466970
Title: Plasmablast Detection From IgG4-Related Disease Patients
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Meir Medical Center (Other)
Responsible Party: Principal Investigator, yair levy, head of internal medicin E, Meir Medical Center
Other Study IDs: 0217-17
Record Dates: First submitted 2018-02-25; First posted 2018-03-15 (Actual); Last update posted 2018-03-16 (Actual); Status verified 2018-03

CONDITIONS: IgG4-related Disease
MeSH Terms: conditions — Immunoglobulin G4-Related Disease

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — 20 samples of IgG4 patients and 20 healthy donors
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- IgG4 patient: 20 samples of IgG4 patients
- healthy donors: 20 healthy donors

SUMMARY:
IgG4-related disease (IgG4-RD) is an immune-mediated, fibro-inflammatory disease that leads to tissue damage, organ dysfunction and, if untreated, to organ failure. The disease can affect almost any anatomic location, but the sites involved most commonly are the pancreas, salivary glands, orbital adnexa, lymph nodes, and retroperitoneum. IgG4-RD, typically diagnosed among individuals who are middle-aged, is characterized by a male predominance except with regard to organs of the head and neck (e.g., the salivary glands and orbits), where the gender distribution is approximately equal. The epidemiology of IgG4-RD remains poorly understood because of its recognition only recently as a multi-organ disease. However, IgG4-RD accounts for many conditions once regarded as disparate, single-organ disorders The purpose of our study is to evaluate the method of plasmablast measurement in peripheral blood of IgG4-RD patients, for diagnosis and follow-up on disease progression and response to treatment. This document will outline the collection, processing and testing procedures for measuring plasmablasts from IgG4-RD patients

DETAILED DESCRIPTION:
IgG4-related disease (IgG4-RD) is an immune-mediated, fibro-inflammatory disease that leads to tissue damage, organ dysfunction and, if untreated, to organ failure. The disease can affect almost any anatomic location, but the sites involved most commonly are the pancreas, salivary glands, orbital adnexa, lymph nodes, and retroperitoneum. IgG4-RD, typically diagnosed among individuals who are middle-aged, is characterized by a male predominance except with regard to organs of the head and neck (e.g., the salivary glands and orbits), where the gender distribution is approximately equal. The epidemiology of IgG4-RD remains poorly understood because of its recognition only recently as a multi-organ disease. However, IgG4-RD accounts for many conditions once regarded as disparate, single-organ disorders.

The current gold standard for the diagnosis of IgG4-RD is the identification of characteristic histology and immunohistochemistry features through biopsy. These pathology features are consistent across the full range of organs affected by IgG4-RD. However, histopathologic variation can occur according to the stage of the lesion; that is, longstanding disease may be predominately fibrotic and a cellular. Confirming the diagnosis of IgG4-RD in such cases can be difficult. Moreover, IgG4-RD organ pathology and IgG4-RD mimickers, such as granulomatosis with polyangiitis (formerly Wegener's), sarcoidosis, histiocytosis, and malignancies (e.g., lymphoma and adenocarcinoma of the pancreas), may share similar features including an IgG4-positive plasma cell infiltrate. Reliance upon serum IgG4 concentrations to diagnose IgG4-RD is similarly problematic because both the specificity and positive predictive value of serum IgG4 concentrations are poor.

Plasmablasts, derived from the B-cell lineage and characterized as CD19lowCD20-CD38+CD27+, comprise a stage intermediate between activated B-cells and plasma cells. Plasmablasts are generally rare in the peripheral blood of healthy individuals, but expansions are observed briefly during responses to infection or vaccination. In contrast, in the setting of autoimmunity and persistent self-antigen(s), plasmablasts can circulate for prolonged periods.

Circulating plasmablasts have been described previously in inflammatory bowel disease, rheumatoid arthritis, systemic lupus erythematosus, and multiple myeloma. Recently, several studies identified plasmablsts in IgG4-RD both as a diagnostic tool and as an indicator of response to treatment

2. Aim

The purpose of our study is to evaluate the method of plasmablast measurement in peripheral blood of IgG4-RD patients, for diagnosis and follow-up on disease progression and response to treatment. This document will outline the collection, processing and testing procedures for measuring plasmablasts from IgG4-RD patients.

3. Plasmablast source

Plasmablasts will be isolated from peripheral blood derived from patients and normal donors who consent to participate in the study. Blood samples will be drawn by a physician or accredited nurse, transferred to the research lab in order to separate PMBCs, which will be stained for CD19lowCD20-CD38+CD27+ markers and measured by flow cytometry (FACS) located at the hematology lab

ELIGIBILITY:
Inclusion Criteria:

1. Patients that obtaining their written consent.
2. Patients above the age of 18 and referred to the Rheumatology clinic or Internal Medicine E Department at the Meir Medical Center for investigation or treatment of IgG4-RD will be candidates to participate in the study.
3. Patients at their primary diagnosis or follow up will be eligible for this study.

Exclusion Criteria:

1. Patient that not diagnosed before with IgG4.
2. patients that does not referred to the Rheumatology clinic or Internal Medicine E Department at the Meir Medical Center.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: There will be 2 groups in the study. One group of 20 IgG4 patients and the other group is 20 healthy donors.
Sampling Method: Non-Probability Sample
Enrollment: 40 (Estimated)
Dates: Start 2018-04-01 (Estimated); Primary Completion 2019-03-01 (Estimated); Study Completion 2019-04-01 (Estimated)

PRIMARY OUTCOMES:
plasmablast measurement in peripheral blood of IgG4-RD patients | 1 year
  Plasmablasts will be isolated from peripheral blood derived from patients and normal donors who consent to participate in the study. Blood samples will be drawn by a physician or accredited nurse, transferred to the research lab in order to separate PMBCs, which will be stained for CD19lowCD20-CD38+CD27+ markers and measured by flow cytometry (FACS) located at the hematology lab.

CONTACTS AND LOCATIONS:
Overall Officials: Yair Levy, prof, Principal Investigator — head of internal medicin E
Locations (2):
- Israel (2):
  - Yael Eizikovits, Kfar Saba
  - Meir health center, Kfar Saba